CLINICAL TRIAL: NCT07073612
Title: Transcatheter Fontan Stenting: Impact on Hepatic Stiffness and Exercise Capacity
Status: Recruiting | Type: Observational
Sponsor: Children's Hospital Los Angeles (Other)
Responsible Party: Principal Investigator, Neil Patel, Medical Staff/USC Faculty CWR • Cardiology CWR, Children's Hospital Los Angeles
Other Study IDs: CHLA-25-00052
Record Dates: First submitted 2025-07-10; First posted 2025-07-18 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: Single-ventricle; Stenosis
Keywords: Stent; fontan; Single-ventricle
MeSH Terms: conditions — Univentricular Heart; Constriction, Pathologic | interventions — Exercise Test

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Cohort: Single ventricle fontan.
  Interventions: Diagnostic Test: Cardiopulmonary Exercise Testing (CPET); Diagnostic Test: Shear Wave Elastography Scan

INTERVENTIONS:
Diagnostic Test: Cardiopulmonary Exercise Testing (CPET) — CPET will be performed on a cycle ergometer using a ramp protocol designed to achieve an exercise time of 8-12 min. The entire procedure duration is approximately 60 min. CPET will be completed 6 months to 1 day before the cardiac catheterization and will be repeated 3-6 months following cardiac catheterization.
Diagnostic Test: Shear Wave Elastography Scan — The study lasts approximately 20 minutes. Shear Wave Elastography will be completed 6 months to 1 day before the cardiac catheterization. The Scan will be repeated 2-4 weeks following cardiac catheterization, and 3-6 months following cardiac catheterization.

SUMMARY:
The goal of this observational study is to assess the clinical impact following Fontan stent placement for extracardiac Fontan conduit (EFC) stenosis in patients with single-ventricle Fontan-palliated patients ages 12-21 years old.

The main question it aims to:

-Assess changes in exercise capacity by cardiopulmonary exercise testing and liver stiffness assessed by shear wave elastography before and after EFC stenting.

Participants will undergo two cardiopulmonary exercise tests and three shear wave elastography scans.

ELIGIBILITY:
Inclusion Criteria:

* Functionally single-ventricle Fontan-palliated patients undergoing clinically indicated cardiac catheterization
* Anticipated Fontan stent placement for extracardiac Fontan conduit stenosis at the discretion of the primary operator
* Weight ≥ 50 kg
* 12-21 years of age

Exclusion Criteria:

* Interrupted IVC
* Greater than mild atrioventricular valve regurgitation on most recent echocardiogram or MRI (RF > 20%).
* Greater than mild systemic ventricular dysfunction on most recent echo or MRI (EF < 40%).
* Non-sinus rhythm
* Pacemaker
* Inability to perform exercise test due to developmental or physical disability

Ages: 12 Years to 21 Years | Sex: All
Age Groups: Child, Adult
Study Population: Patients 12-21 years old with functioning single-ventricle Fontan-palliated who are scheduled to undergo clinically indicated fontan conduit stenting.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2027-12-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Determine change from baseline in exercise capacity after Fontan stenting. | 1 year post enrollment
  Peak oxygen consumption (VO2) as measured by Vyntus CPX metabolic cart.
Determine changes from baseline in liver stiffness as measured by shear wave elastography after Fontan stenting. | 1 year post enrollment
  FibroScan will be used to assess liver stiffness before catheterization, at 2-4 weeks following stent placement, and 3-6 months following stent placement.

CONTACTS AND LOCATIONS:
Overall Officials: Neil Patel, MD, Principal Investigator — Children's Hospital Los Angeles
Locations (1):
- Children's Hospital Los Angeles, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No